CLINICAL TRIAL: NCT05041257
Title: A Phase 2, Single Arm Study of Mirvetuximab Soravtansine in Recurrent Platinum-Sensitive, High-Grade Epithelial Ovarian, Primary Peritoneal, or Fallopian Tube Cancers With High Folate Receptor-Alpha Expression
Brief Title: Mirvetuximab Soravtansine Monotherapy in Platinum-Sensitive Epithelial, Peritoneal, and Fallopian Tube Cancers
Acronym: PICCOLO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IMGN853-0419; 2021-003592-34 (EudraCT Number)
Record Dates: First submitted 2021-08-24; First posted 2021-09-13 (Actual); Results first posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Ovarian Cancer; Peritoneal Cancer; Fallopian Tube Cancer
Keywords: Platinum-sensitive; Ovarian cancer; Folate-receptor alpha expression; Antibody-drug conjugate; Cancer; Ovarian Neoplasma; Recurrent Platinum-Sensitive; High-Grade Ovarian; PICCOLO
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms; Neoplasms | interventions — mirvetuximab soravtansine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Mirvetuximab Soravtansine (Experimental): Participants will receive MIRV 6.0 mg/kg adjusted by ideal body weight (AIBW)
  Interventions: Drug: Mirvetuximab soravtansine

INTERVENTIONS:
Drug: Mirvetuximab soravtansine — Administered by intravenous (IV) infusion on Day 1 of every 3-week cycle
  Other Names: MIRV; IMGN853

SUMMARY:
PICCOLO (IMGN853-0419) is a Phase 2 multicenter, open label study designed to evaluate the safety and efficacy of Mirvetuximab Soravtansine in participants with platinum-sensitive ovarian, primary peritoneal or fallopian tube cancers with high folate receptor-alpha (FRα) expression.

DETAILED DESCRIPTION:
Mirvetuximab Soravtansine (MIRV) is an investigational antibody drug conjugate designed to selectively kill cancer cells. The antibody (protein) part of MIRV targets tumors by delivering a cell-killing drug to the tumor cells carrying a tumor-associated protein called folate receptor alpha (FRα). It is being developed for the treatment of participants with recurrent platinum-sensitive, high-grade epithelial ovarian, primary peritoneal, or fallopian tube cancers with high folate receptor-alpha expression. Participants will have had at least 2 prior lines of therapy. These will include at least 2 lines of platinum-containing therapy or 1 line with a documented platinum allergy. FRα positivity will be defined by the Ventana FOLR1 (FOLR1- 2.1) CDx assay (Ventana FOLR1 Assay).

ELIGIBILITY:
Inclusion Criteria:

1. Participants ≥ 18 years of age
2. Participants must have an Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0 or 1
3. Participants must have a confirmed diagnosis of high-grade serous epithelial ovarian cancer (EOC), primary peritoneal cancer, or fallopian tube cancer
4. Participants must have platinum-sensitive disease defined as radiographic progression greater than 6 months from last dose of most recent platinum therapy Note: Progression should be calculated from the date of the last administered dose of platinum therapy to the date of the radiographic imaging showing progression
5. Participants must have progressed radiographically on or after their most recent line of anticancer therapy
6. Participants must have at least 1 lesion that meets the definition of measurable disease by Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) (radiologically measured by the Investigator)
7. Participants must be willing to provide an archival tumor tissue block or slides, or undergo procedure to obtain a new biopsy using a low-risk, medically routine procedure for immunohistochemistry (IHC) confirmation of FRα positivity
8. Participant's tumor must be positive for FRα expression as defined by the Ventana FOLR1 Assay
9. Prior anticancer therapy

   1. Participants must have received at least 2 prior systemic lines of platinum therapy and be considered by the Investigator as appropriate for single-agent non-platinum therapy (documentation required - for example, high risk of hypersensitivity reaction; risk of further cumulative toxicity with additional platinum, including but not limited to myelosuppression, neuropathy, renal insufficiency or other) i. Note: Participants who have had a documented platinum allergy may have had only 1 prior line of platinum
   2. Participants may have received up to but no more than 1 prior independent non-platinum cytotoxic therapy
   3. Participants must have had testing for breast cancer susceptibility gene (BRCA) mutation (tumor or germline) and, if positive, must have received a prior poly (ADP-ribose) polymerase (PARP) inhibitor as either treatment or maintenance therapy
   4. Neoadjuvant ± adjuvant therapies are considered 1 line of therapy
   5. Maintenance therapy (for example, bevacizumab, PARP inhibitors) will be considered part of the preceding line of therapy (that is, not counted independently)
   6. Therapy changed due to toxicity in the absence of progression will be considered part of the same line (that is, not counted independently)
10. Participants must have completed prior therapy within the specified times below:

    1. Systemic antineoplastic therapy within 5 half-lives or 4 weeks (whichever is shorter) prior to first dose of MIRV
    2. Focal radiation completed at least 2 weeks prior to first dose of MIRV
11. Participants must have stabilized or recovered (Grade 1 or baseline) from all prior therapy-related toxicities (except alopecia)
12. Participants must have completed any major surgery at least 4 weeks prior to first dose of MIRV and have recovered or stabilized from the side effects of prior surgery prior to first dose of MIRV
13. Participants must have adequate hematologic, liver and kidney functions defined as:

    1. Absolute neutrophil count (ANC) ≥ 1.5 x 10^9/liter (L) (1500/microliter [μL]) without granulocyte colony-stimulating factor (G-CSF) in the prior 10 days or long-acting white blood cell (WBC) growth factors in the prior 20 days
    2. Platelet count ≥ 100 x 10^9/L (100,000/μL) without platelet transfusion in the prior 10 days
    3. Hemoglobin ≥ 9.0 grams (g)/deciliter (dL) without packed red blood cell (PRBC) transfusion in the prior 21 days
    4. Serum creatinine ≤ 1.5 x upper limit of normal (ULN)
    5. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3.0 x ULN
    6. Serum bilirubin ≤ 1.5 x ULN (participants with documented diagnosis of Gilbert syndrome are eligible if total bilirubin < 3.0 x ULN)
    7. Serum albumin ≥ 2 g/dL
14. Participants must be willing and able to sign the informed consent form (ICF) and to adhere to the protocol requirements
15. Women of childbearing potential (WCBP) must agree to use highly effective contraceptive method(s) while on MIRV and for at least 3 months after the last dose
16. WCBP must have a negative pregnancy test within the 4 days prior to the first dose of MIRV

Exclusion Criteria:

1. Participants with endometrioid, clear cell, mucinous, or sarcomatous histology, mixed tumors containing any of the above histologies, or low-grade/ borderline ovarian tumor
2. Participants with prior wide-field radiotherapy (RT) affecting at least 20% of the bone marrow
3. Participants with > Grade 1 peripheral neuropathy per Common Terminology Criteria for Adverse Events (CTCAE)
4. Participants with active or chronic corneal disorders, history of corneal transplantation, or active ocular conditions requiring ongoing treatment/monitoring, such as uncontrolled glaucoma, wet age-related macular degeneration requiring intravitreal injections, active diabetic retinopathy with macular edema, macular degeneration, presence of papilledema, and/or monocular vision
5. Participants with serious concurrent illness or clinically relevant active infection, including, but not limited to the following:

   1. Active hepatitis B or C infection (whether or not on active antiviral therapy)
   2. Human immunodeficiency virus (HIV) infection
   3. Active cytomegalovirus infection
   4. Any other concurrent infectious disease requiring IV antibiotics within 2 weeks prior to the first dose of MIRV

   Note: Testing at screening is not required for the above infections unless clinically indicated.
6. Participants with a history of multiple sclerosis (MS) or other demyelinating disease and/or Lambert-Eaton syndrome (paraneoplastic syndrome)
7. Participants with clinically significant cardiac disease including, but not limited to, any of the following:

   1. Myocardial infarction ≤ 6 months prior to first dose
   2. Unstable angina pectoris
   3. Uncontrolled congestive heart failure (New York Heart Association > class II)
   4. Uncontrolled ≥ Grade 3 hypertension (per CTCAE)
   5. Uncontrolled cardiac arrhythmias
8. Participants with a history of hemorrhagic or ischemic stroke within 6 months prior to enrollment
9. Participants with a history of cirrhotic liver disease (Child-Pugh Class B or C)
10. Participants with a previous clinical diagnosis of noninfectious interstitial lung disease (ILD), including noninfectious pneumonitis
11. Participants requiring use of folate-containing supplements (for example, folate deficiency)
12. Participants with prior hypersensitivity to monoclonal antibodies (mAb)
13. Women who are pregnant or breastfeeding
14. Participants who received prior treatment with MIRV or other FRα-targeting agents
15. Participants with untreated or symptomatic central nervous system (CNS) metastases
16. Participants with a history of other malignancy within 3 years prior to enrollment

    Note: Participants with tumors with a negligible risk for metastasis or death (for example, adequately controlled basal-cell carcinoma or squamous-cell carcinoma of the skin, or carcinoma in situ of the cervix or breast) are eligible.
17. Prior known hypersensitivity reactions to study drugs and/or any of their excipients

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2021-10-19 (Actual); Primary Completion 2024-12-12 (Actual); Study Completion 2024-12-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (35):
- United States (11):
  - City of Hope National Medical Center /ID# 269928, Duarte, California
  - University of California Los Angeles /ID# 269969, Los Angeles, California
  - University Colorado Cancer Center /ID# 269930, Aurora, Colorado
  - Women'S Cancer Care /ID# 269925, Covington, Louisiana
  - Holy Name Medical Center /ID# 269927, Teaneck, New Jersey
  - Cleveland Clinic Main Campus /ID# 269922, Cleveland, Ohio
  - The Mark H Zangmeister Center /ID# 269929, Columbus, Ohio
  - Women & Infants Hospital /ID# 269923, Providence, Rhode Island
  - Duplicate_SCRI - Tennessee Oncology /ID# 269921, Nashville, Tennessee
  - Texas Oncology - South Austin /ID# 269924, Austin, Texas
  - Virginia Oncology Associates - Norfolk (Lake Wright) /ID# 269926, Norfolk, Virginia
- Australia (2):
  - Newcastle Private Hosptial /ID# 269734, Lambton Heights, New South Wales
  - Monash Health - Monash Medical Centre /ID# 269735, Clayton, Victoria
- Belgium (3):
  - UZ Gent /ID# 269737, Ghent, Oost-Vlaanderen
  - Universitair Ziekenhuis Leuven /ID# 269736, Leuven, Vlaams-Brabant
  - UCL Namur University Hospital, Site Sainte-Elisabeth /ID# 269738, Namur
- France (4):
  - Centre Armoricain de Radiotherapie Imagerie & Oncologie (CARIO) /ID# 269847, Plérin, Cotes-d Armor
  - Institut de Cancérologie de l'Ouest René Gauducheau /ID# 269846, Saint-Herblain, Loire-Atlantique
  - Centre Leon Berard /ID# 269848, Lyon, Rhone
  - Institut de cancérologie Strasbourg Europe (ICANS) /ID# 269849, Strasbourg
- Ireland (2):
  - Bon Secours Cork Hospital /ID# 269851, Cork
  - Waterford Regional Hospital /ID# 269852, Waterford
- Italy (5):
  - Istituto Nazionale Dei Tumori /ID# 269864, Milan, Milano
  - Istituto Europeo Di Oncologia /ID# 269860, Milan, Milano
  - Istituto Nazionale Tumori Irccs Fondazione G. Pascale /ID# 269863, Naples, Napoli
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS-Università Cattolica /ID# 269861, Rome, Roma
  - IRCCS AOU di Bologna Policlinico Sant Orsola Malpighi /ID# 269862, Bologna
- Spain (8):
  - Hospital Universitario Reina Sofia /ID# 269892, Córdoba, Cordoba
  - Hospital Universitario de Jaén /ID# 269895, Jaén, Jaen
  - Hospital Universitario Vall d'Hebron /ID# 269889, Barcelona
  - Hospital MD Anderson Cancer Center Madrid /ID# 269888, Madrid
  - Hospital Universitario La Paz /ID# 269890, Madrid
  - Hospital Universitario HM Sanchinarro /ID# 269891, Madrid
  - Hospital Universitario Virgen del Rocio /ID# 269894, Seville
  - Hospital Clínico Universitario de Valencia /ID# 269893, Valencia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Alvarez Secord A, Lewin SN, Murphy CG, Cecere SC, Barquin A, Galvez-Montosa F, Mathews CA, Konecny GE, Ray-Coquard I, Oaknin A, Rubio Perez MJ, Bonaventura A, Diver EJ, Ayuk SM, Wang Y, Corr BR, Salutari V. The efficacy and safety of mirvetuximab soravtansine in FRalpha-positive, third-line and later, recurrent platinum-sensitive ovarian cancer: the single-arm phase II PICCOLO trial. Ann Oncol. 2025 Mar;36(3):321-330. doi: 10.1016/j.annonc.2024.11.011. Epub 2024 Nov 29. PMID 39617145
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=IMGN853-0419

RESULTS

PARTICIPANT FLOW:
Groups:
- Mirvetuximab Soravtansine: Participants received single-agent mirvetuximab soravtansine at 6 milligrams (mg)/kilogram (kg) adjusted by ideal body weight (AIBW) administered through intravenous (IV) infusion on Day 1 of every 3-week cycle.
Period: Overall Study
Arm/Group | Mirvetuximab Soravtansine
Started | 79
Received at Least 1 Dose of Study Drug | 79
Completed | 0
Not Completed | 79
Not completed — Death | 37
Not completed — Lost to Follow-up | 3
Not completed — Sponsor decision | 39

BASELINE CHARACTERISTICS:
Population: Safety Population included all participants who received at least 1 dose of mirvetuximab soravtansine.
Groups:
- Mirvetuximab Soravtansine: Participants received single-agent mirvetuximab soravtansine at 6 mg/kg AIBW administered through IV infusion on Day 1 of every 3-week cycle.
Arm/Group | Mirvetuximab Soravtansine
Number analyzed (Participants) | 79
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.1 (10.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 79
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 68
  Unknown or Not Reported | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 65
  More than one race | 0
  Unknown or Not Reported | 9

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) Assessed by Investigator Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1])
Description: ORR was defined as percentage of participants with a confirmed best overall response (BOR) of complete response (CR) or partial response (PR). CR: Disappearance of all target or non-target lesions. All pathological or non-pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 millimeters (mm). PR: At least 30% decrease in the sum of the longest diameters (SoD) of target lesions, taking as reference the baseline SoD.
Time Frame: Up to 3 years
Population: Efficacy Evaluable Population Per Investigator included all participants who received at least 1 dose of mirvetuximab soravtansine and had measurable disease at baseline per Investigator.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Mirvetuximab Soravtansine
Number analyzed (Participants) | 79
percentage of participants | 51.9 [40.4 to 63.3]

2. Secondary Outcome: Duration of Response (DOR) Assessed by the Investigator Using RECIST v1.1
Description: DOR was defined as the time from the date of the first response (CR or PR), until the date of progressive disease (PD) or death from any cause, whichever occurred first. DOR for participants who had not progressed or died at the time of analysis was censored at the date of their last tumor assessment. PD: At least a 20% increase in the SoD of target lesion, taken as reference the smallest (nadir) SoD since and including baseline. In addition to the relative increase of 20%, the SoD must also demonstrate an absolute increase of at least 5 mm. Unequivocal progression of non-target lesions. Unequivocal progression should not normally trump target lesion status. It must be representative of overall disease status change, not a single lesion increase. DOR was estimated using the Kaplan-Meier method.
Time Frame: Up to 3 years
Population: Efficacy Evaluable Population Per Investigator included all participants who received at least 1 dose of mirvetuximab soravtansine and had measurable disease at baseline per Investigator. 'Overall number of participants analyzed' = participants with objective response.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Mirvetuximab Soravtansine
Number analyzed (Participants) | 41
months | 8.25 [5.55 to 10.78]

3. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was defined as any untoward medical occurrence that developed or worsened in severity during the conduct of a clinical study and does not necessarily had a causal relationship to study drug. TEAEs were defined as AEs with an onset date on or after the first dose of Study drug, and within 30 days of the last dose of study drug or prior to the start of a new anticancer treatment, whichever occurred first. A summary of all Serious Adverse Events (SAEs) and Other Adverse Events (nonserious) regardless of causality is located in the 'Reported Adverse Events' Section.
Time Frame: Up to 3 years
Population: Safety Population included all participants who received at least 1 dose of mirvetuximab soravtansine.
Measure: Count of Participants; unit: Participants
Arm/Group | Mirvetuximab Soravtansine
Number analyzed (Participants) | 79
Participants | 78

4. Secondary Outcome: Percentage of Participants With CA-125 Confirmed Clinical Response Per Gynecologic Cancer Intergroup (GCIG) Criteria
Description: The GCIG CA-125 response was defined as at least 50% reduction in CA-125 levels from baseline. The response must have been confirmed and maintained for at least 28 days.
Time Frame: Up to 3 years
Population: CA-125 Response-Evaluable Population included all participants who received at least 1 dose of mirvetuximab soravtansine, whose pretreatment sample was ≥ 2.0 times the upper limit of normal (ULN), within 2 weeks prior to first dose of mirvetuximab soravtansine, and who had at least 1 post-baseline CA-125 evaluation.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Mirvetuximab Soravtansine
Number analyzed (Participants) | 47
percentage of participants | 74.5 [59.7 to 86.1]

5. Secondary Outcome: Progression-Free Survival (PFS) as Assessed by the Investigator Using RECIST v1.1
Description: PFS was defined as the time from initiation of study drug until the date of PD or death whichever occurred first, estimated using the Kaplan-Meier method. PD: At least a 20% increase in the SoD of target lesion, taken as reference the smallest (nadir) SoD since and including baseline. In addition to the relative increase of 20%, the SoD must also demonstrate an absolute increase of at least 5 mm. Unequivocal progression of non-target lesions and appearance of new lesions. Unequivocal progression should not normally trump target lesion status. It must be representative of overall disease status change, not a single lesion increase.
Time Frame: Up to 3 years
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Mirvetuximab Soravtansine
Number analyzed (Participants) | 79
months | 6.93 [5.85 to 9.59]

6. Secondary Outcome: Overall Survival Assessed by the Investigator Using RECIST v1.1
Description: Overall survival was defined as the time from the date of first dose until the date of death from any cause, estimated using the Kaplan-Meier method.
Time Frame: Up to 3 years
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Mirvetuximab Soravtansine
Number analyzed (Participants) | 79
months | 27.17 [23.79 to NA] — Due to insufficient number of participants with an event, upper limit of 95% confidence interval (CI) could not be calculated.

ADVERSE EVENTS:
Time Frame: All-cause mortality and adverse event tables include events reported from the start of safety data collection to the end of the study. The median time on follow-up was 26.5 months.
Description: Safety Population included all participants who received at least 1 dose of mirvetuximab soravtansine.
Arm/Group | Mirvetuximab Soravtansine
All-Cause Mortality (participants affected / at risk) | 37/79
Serious Adverse Events (participants affected / at risk) | 17/79
Other Adverse Events (participants affected / at risk) | 77/79
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mirvetuximab Soravtansine (N=79)
KERATITIS (Eye disorders) | 1 (1)
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 1 (1)
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 (2)
SUBILEUS (Gastrointestinal disorders) | 1 (1)
VOMITING (Gastrointestinal disorders) | 1 (1)
EXTRAVASATION (General disorders) | 1 (1)
SUPRAPUBIC PAIN (General disorders) | 1 (1)
CYSTITIS (Infections and infestations) | 1 (1)
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (1)
PNEUMONIA (Infections and infestations) | 1 (1)
PYELONEPHRITIS (Infections and infestations) | 1 (1)
SEPTIC SHOCK (Infections and infestations) | 1 (2)
GASTROINTESTINAL STOMA COMPLICATION (Injury, poisoning and procedural complications) | 1 (1)
ATAXIA (Nervous system disorders) | 1 (1)
NEUROPATHY PERIPHERAL (Nervous system disorders) | 1 (1)
SYNCOPE (Nervous system disorders) | 1 (1)
THROMBOTIC STROKE (Nervous system disorders) | 1 (1)
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 4 (7)
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 1 (1)
DEEP VEIN THROMBOSIS (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mirvetuximab Soravtansine (N=79)
ANAEMIA (Blood and lymphatic system disorders) | 7 (11)
NEUTROPENIA (Blood and lymphatic system disorders) | 11 (34)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 5 (9)
CATARACT (Eye disorders) | 27 (41)
CORNEAL EPITHELIAL MICROCYSTS (Eye disorders) | 5 (11)
DRY EYE (Eye disorders) | 32 (49)
EYE PAIN (Eye disorders) | 5 (9)
KERATITIS (Eye disorders) | 6 (12)
KERATOPATHY (Eye disorders) | 26 (57)
PHOTOPHOBIA (Eye disorders) | 13 (19)
VISION BLURRED (Eye disorders) | 52 (116)
VISUAL ACUITY REDUCED (Eye disorders) | 7 (9)
VITREOUS FLOATERS (Eye disorders) | 6 (6)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 6 (6)
ABDOMINAL PAIN (Gastrointestinal disorders) | 14 (18)
CONSTIPATION (Gastrointestinal disorders) | 14 (17)
DIARRHOEA (Gastrointestinal disorders) | 24 (46)
FLATULENCE (Gastrointestinal disorders) | 4 (5)
NAUSEA (Gastrointestinal disorders) | 29 (42)
STOMATITIS (Gastrointestinal disorders) | 5 (5)
VOMITING (Gastrointestinal disorders) | 14 (18)
ASTHENIA (General disorders) | 24 (40)
FATIGUE (General disorders) | 14 (22)
PYREXIA (General disorders) | 8 (8)
COVID-19 (Infections and infestations) | 13 (13)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 15 (23)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 17 (25)
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 7 (8)
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 4 (5)
WEIGHT DECREASED (Investigations) | 5 (7)
DECREASED APPETITE (Metabolism and nutrition disorders) | 7 (8)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 8 (12)
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 9 (12)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 5 (9)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 19 (24)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 4 (4)
MYALGIA (Musculoskeletal and connective tissue disorders) | 7 (9)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 6 (7)
DIZZINESS (Nervous system disorders) | 4 (5)
DYSGEUSIA (Nervous system disorders) | 9 (10)
HEADACHE (Nervous system disorders) | 13 (18)
NEUROPATHY PERIPHERAL (Nervous system disorders) | 22 (37)
NEUROTOXICITY (Nervous system disorders) | 10 (14)
PARAESTHESIA (Nervous system disorders) | 5 (10)
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 7 (11)
ANXIETY (Psychiatric disorders) | 4 (4)
INSOMNIA (Psychiatric disorders) | 5 (6)
COUGH (Respiratory, thoracic and mediastinal disorders) | 6 (7)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 8 (11)
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 6 (6)
ERYTHEMA (Skin and subcutaneous tissue disorders) | 4 (4)
HYPERTENSION (Vascular disorders) | 4 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2021-12-22): https://cdn.clinicaltrials.gov/large-docs/57/NCT05041257/Prot_000.pdf
  • Statistical Analysis Plan (2024-02-26): https://cdn.clinicaltrials.gov/large-docs/57/NCT05041257/SAP_001.pdf